CLINICAL TRIAL: NCT00944723
Title: Evaluation of the Use of Plasma Zinc Concentration for Assessing the Impact of Targeted and Mass Zinc Fortification Programs
Brief Title: Impact of Mass Zinc Fortification Programs on Plasma Zinc Concentration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Helen Keller International (Other); Cheikh Anta Diop University, Senegal (Other); Global Alliance for Improved Nutrition (Other)
Responsible Party: Prof. Kenneth H. Brown, Helen Keller International
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 107008-2; 200816610
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Zinc Deficiency
Keywords: zinc fortification; zinc supplementation; plasma zinc concentration
MeSH Terms: interventions — Zinc Sulfate; Vitamin B Complex; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Zinc-fortified bread (10 mg zinc/d) (Experimental): Daily consumption of zinc fortified bread for 1 month
  Interventions: Dietary Supplement: Zinc-fortified bread; Dietary Supplement: Placebo supplement
- Zinc fortified bread (20 mg zinc/d) (Experimental): Daily consumption of zinc fortified bread for 1 month.
  Interventions: Dietary Supplement: Zinc-fortified bread; Dietary Supplement: Placebo supplement
- Zinc supplemented group (Experimental): Daily consumption of non-fortified bread and daily intake of zinc supplement (10 mg zinc/d)
  Interventions: Dietary Supplement: Zinc supplement; Dietary Supplement: Non-fortified bread
- Non-fortified group (Placebo Comparator): Daily consumption of non-fortified bread and a placebo supplement for 1 month.
  Interventions: Dietary Supplement: Non-fortified bread; Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Zinc-fortified bread — Bread made with zinc-fortified wheat flour
  Other Names: Les Grands Moulins de Dakar
  Arms: Zinc fortified bread (20 mg zinc/d); Zinc-fortified bread (10 mg zinc/d)
Dietary Supplement: Zinc supplement — Liquid supplement with zinc
  Other Names: Zinc sulfate and B vitamins, DSM
  Arms: Zinc supplemented group
Dietary Supplement: Non-fortified bread — Daily consumption of non-fortified bread
  Other Names: Les Grands Moulins de Dakar
  Arms: Non-fortified group; Zinc supplemented group
Dietary Supplement: Placebo supplement — Daily intake of placebo supplement
  Other Names: B-vitamins, DSM
  Arms: Non-fortified group; Zinc fortified bread (20 mg zinc/d); Zinc-fortified bread (10 mg zinc/d)

SUMMARY:
The purpose of the study is to evaluate the use of plasma zinc concentration for assessing the impact of mass zinc fortification programs.

DETAILED DESCRIPTION:
The objectives of the present study are to determine whether plasma zinc concentration changes in response to additional zinc consumption, as provided by zinc-fortified cereal-based complementary foods fed to adult men (fortified at a level consistent with currently proposed levels). The following specific steps will be completed:

1. Zinc-fortified breads prepared from zinc-fortified wheat flour will be developed with assistance from experts in food technology.
2. A four-week feeding trial will be implemented to assess the change in plasma zinc concentration among young adult men who receive: a) bread fortified with a moderate amount of zinc and a liquid vitamin preparation between meals; b) bread fortified with a large amount zinc and a liquid vitamin preparation between meals; c) non-zinc-fortified bread and a liquid vitamin preparation between meals [negative control group]; and d) non-zinc-fortified bread and a zinc-containing liquid vitamin preparation between meals [positive control group].

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy males

Exclusion Criteria:

* Hemoglobin <80 g/L

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Plasma zinc concentration | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Brown, MD, Principal Investigator — University of California, Davis
Locations (1):
- Helen Keller International, Dakar, Senegal

REFERENCES:
- [Derived] Aaron GJ, Ba Lo N, Hess SY, Guiro AT, Wade S, Brown KH. Plasma zinc concentration increases within 2 weeks in healthy Senegalese men given liquid supplemental zinc, but not zinc-fortified wheat bread. J Nutr. 2011 Jul;141(7):1369-74. doi: 10.3945/jn.110.136952. Epub 2011 May 11. PMID 21562238